CLINICAL TRIAL: NCT02064699
Title: Assessing the Risk of CMV Infection of the Renal Transplant About R + by Cellular Immunity Analyzed by the QuantiFERON ®-CMV Test.
Acronym: QUANTIC-R+
Status: Terminated | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I10002 QUANTIC-R+
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Renal Transplant Recipient; Immunized Against the Cytomegalovirus
Keywords: Renal transplant; CMV; Test QuantiFERON-CMV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Detection of the CMV in sang, the leukocytes, or plasma with or without the viral quantification.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CMV infection: Renal transplant recipient immunized against the Cytomegalovirus
  Interventions: Biological: CMV Infection

INTERVENTIONS:
Biological: CMV Infection — Routine follow-up (viral load, creatininaemia, neutrophil count, isolation of CMV strains when possible) and biological sample collection for.
  Using the QuantiFERON-CMV test for predicting the risk of CMV infection in the transplanted immune against CMV.

SUMMARY:
Cytomegalovirus (CMV) infection was observed in over 30% of organ recipients with high morbidity. Moreover, no prophylaxis, 75% R + D-transplanted, 55%, R + D + and D-25% R + develop CMV. The number of available antiviral drugs is reduced and noticeable side effects (neutropenia, renal toxicity) lead to premature discontinuation of therapy or the use of reduced doses that promote non-response to treatment and the emergence of resistance. In case of neutropenia, there are more an increased risk of secondary rejection due to the reduction of immunosuppressive treatment rendered necessary by the haematological reached.

Rational use of these molecules is necessary with essential today as the optimal duration of prophylaxis primary issues and the prophylaxis of recurrences in case of CMV infection reported in.

DETAILED DESCRIPTION:
QuantiFERON-CMV ® is a fast and standardized test that evaluates the CMV specific cellular immunity measuring the amount of secreted Interferon gamma (IFN gamma) in plasma by ELISA. It uses more epitopes of proteins including CMV glycoprotein B (gB), protein IE-1 and protein pp65 and protein pp50, which are specific for (human leukocyte antigen) HLA class I. Pretreatment of the sample is simple and plasma can be stored, frozen, for a delayed dose of interferon.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipient
* Immunized against the Cytomegalovirus

Exclusion Criteria:

* Not willing to participate, no health insurance
* clinical evidence of active viral infection
* renal transplant recipient whose treatment includes induction antilymphocyte antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipient Immunized against the Cytomegalovirus.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Predictive values of Cytomegalovirus infection | 1 week
  CMV infection defined by a positive ADNémie confirmed on a second sample ideally one week apart.

SECONDARY OUTCOMES:
No response to treatment | 21 days
  Persistence of an active CMV infection defined by a persistent ADNémie for more than 21 days under antiviral treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie ALAIN, MD, Principal Investigator — Limoges UH
Locations (12):
- France (12):
  - Virologie, Besançon
  - Virologie, Caen
  - Virologie, Clermont-Ferrand
  - Virologie, Grenoble
  - Virologie, Lille
  - Bactériologie Virologie, Limoges
  - Virologie, Nantes
  - Virologie, Reims
  - Virologie, Rennes
  - Virologie, Saint-Etienne
  - Virologie, Strasbourg
  - Foch Hospital, Suresnes

REFERENCES:
- [Background] Rutkow IM. Crawford Williamson Long. Arch Surg. 1999 May;134(5):578. doi: 10.1001/archsurg.134.5.578. No abstract available. PMID 10323437
- [Derived] Mafi S, Essig M, Rerolle JP, Lagathu G, Crochette R, Brodard V, Schvartz B, Gouarin S, Bouvier N, Engelmann I, Garstka A, Bressollette-Bodin C, Cantarovitch D, Germi R, Janbon B, Archimbaut C, Heng AE, Garnier F, Gomes-Mayeras M, Labrunie A, Hantz S, Alain S. Torque teno virus viremia and QuantiFERON(R)-CMV assay in prediction of cytomegalovirus reactivation in R+ kidney transplant recipients. Front Med (Lausanne). 2023 Jun 22;10:1180769. doi: 10.3389/fmed.2023.1180769. eCollection 2023. PMID 37425298